CLINICAL TRIAL: NCT01664832
Title: Is Synchronization More Effective During Noninvasive Ventilation in Immediately Extubated Preterm Infants?
Acronym: N_SIMV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Prof. Dr. Helmut Hummler (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. Helmut Hummler, Prof. Dr. Helmut Hummler, University of Ulm
Organization: University of Ulm (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: ULMN_SIMV
Record Dates: First submitted 2012-08-02; First posted 2012-08-14 (Estimated); Last update posted 2013-06-27 (Estimated); Status verified 2013-06

CONDITIONS: Respiratory Distress Syndrome
Keywords: Premature Infants; snychronized ventilation; non-invasive ventilation; RDS
MeSH Terms: conditions — Respiratory Distress Syndrome; Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- S-nIMV (Experimental): nIMV synchronized using abdominal pressure capsule sensor device
  Interventions: Device: S-nIMV
- nIMV (Placebo Comparator): non-synchronized nasal intermittent mandatory ventilation group
  Interventions: Device: S-nIMV

INTERVENTIONS:
Device: S-nIMV — Synchronization of nasal breaths to infant's own respiratory effort

SUMMARY:
The purpose of this study is the examination of the hypothesis that synchronized nasal IMV as compared to non-synchronized nasal IMV will decrease breathing effort in preterm infants immediately after extubation when recovering from Respiratory distress syndrome (RDS).

Another objective is to examine the effects for synchronized non-invasive mechanical ventilation on gas exchange and cerebral oxygen saturation.

DETAILED DESCRIPTION:
In this study the investigators plan to test the hypothesis that synchronized nasal IMV (S-NIMV) as compared to non-synchronized nasal IMV (NIMV) will decrease breathing effort in preterm infants immediately after extubation when recovery from RDS, as measured by phasic esophageal pressure deflection.

Furthermore, the investigators plan to evaluate the effects of synchronized NIMV on gas exchange and brain oxygenation, and to evaluate the reliability of a newly developed abdominal pressure sensor device for the S-NIMV mode in a newly designed commercially available ventilator device.

ELIGIBILITY:
Inclusion Criteria:

Preterm infants recovering from respiratory failure with the following criteria were eligible for this study.

* Gestational age <32 wks, those who are on invasive mechanical ventilation, recovering from RDS, and ready for extubation as judged by the clinical team.
* Informed consent available.

Exclusion Criteria:

• Infants with major congenital anomalies involving the CNS, lung (i.e. lung hypoplasia, active air leaks) or the heart (ASD, VSD allowed), or known neuromuscular disease.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2012-07; Primary Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
phasic esophageal pressure deflection | 4 hours

SECONDARY OUTCOMES:
Cerebral oxygen saturation | 4 hours
Arterial oxygen saturation | 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Hummler Helmut, Prof. Dr, Principal Investigator — University of Ulm
Locations (1):
- Children's Hospital University of Ulm, Ulm, Baden-Wüttemberg, Germany